CLINICAL TRIAL: NCT04511832
Title: Comparative Effectiveness of Acupuncture and Nonsteroidal Anti-inflammatory Drugs for the Management of Aromatase Inhibitor Induced Arthralgia Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CMUH106-REC3-137
Record Dates: First submitted 2020-07-24; First posted 2020-08-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Acupuncture
MeSH Terms: conditions — Breast Neoplasms | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture to NSAIDs (Experimental)
  Interventions: Drug: Diclofenac
- NSAIDs to Acupuncture (Experimental)
  Interventions: Drug: Diclofenac
- Combined both acupuncture and NSAIDs (Experimental)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac — Patients who were diagnosed as breast cancer and met the inclusion criteria will be recruited and randomly assigned to acupuncture group or drug (NSAIDs) group. After each subgroup completing the 4 weeks intervention, all the participants were enter washout period lasting 2 weeks to eliminate the effect of the previous treatment. Crossover was held after washout period and made the patients to have the other treatment in the following 4 weeks. After receiving the case, the third group recorded the pain indicators for the first month, followed by a one-month trial- combination of acupuncture and NSAID treatment, and then followed up for another month after stopping.

SUMMARY:
Hormone therapy is used to treat women with hormone receptor-positive breast cancer and aromatase inhibitor (AI) is administered after menopause. AI therapy has been proven to be effective in improving the disease-free survival rate, decreasing the recurrence rates and a lower incidence of contralateral breast cancer. However, arthralgia frequently reported as an important adverse event of AI therapy and sometimes resulted in noncompliance with AI therapy. The prevalence of AI induced arthralgia rates ranged from 20 to 74%. Inadequately managed AI induced arthralgia remains a major unmet need in oncology practice in breast cancer survivors.

The goal of this project is to conduct a crossover designed pragmatic clinical trial to evaluate the effectiveness of acupuncture versus NSAID (Diclofenac) for the management of aromatase inhibitor induced arthralgia.

The third group was set to use non-steroidal analgesics plus acupuncture to evaluate the effectiveness of joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Women who were postmenopausal aged more than 20 years old.
* history of stage 0 to III hormone receptor-positive breast cancer, and currently taking a third-generation AI (anastrozole, letrozole, or exemestane) for at least 3 month.
* Those who reported pain and/or stiffness in one or more joints, which started or worsened after initiation of AI therapy had worst joint pain rated at least three or greater on a 0-10 numerical rating scale in the preceding week.

Exclusion Criteria:

* any prior acupuncture use for AI-induced joint symptoms or acupuncture within 1 months before entry
* inflammatory, metabolic, or neuropathic arthropathies
* bone fracture/surgery of an afflicted extremity during the preceding 6 months
* allergy to NSAID
* current use of narcotics
* bleeding or coagulation disorders
* localized skin infections
* needle phobia
* intra-articular corticosteroid within 4 weeks preceding the study
* any severe chronic or uncontrolled comorbid disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Acupuncture can improve joint symptoms resulting from aromatase inhibitor and quality of life | one year
  Patients will be asked to complete a baseline questionnaire covering demographic information and reproductive history. At baseline and at 4, 6 and 10 weeks, self-administered questionnaires including the 10mm visual analogue scales. Follow-up assessments will be conducted at the 4 weeks after the end of intervention.
  According to statistically estimation, we compare the changes between three subgroups and hypothesize 20% difference as significant effect after intervention. We use ANOVA to calculate the sample size with an alpha of 0.05 as significance level, approximately 80% power and 20% drop-out rate. The trial will enroll 145 participants.

CONTACTS AND LOCATIONS:
Overall Officials: China Medicine University China Medicine University, Study Chair — China Medicine University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan